CLINICAL TRIAL: NCT03873961
Title: Short and Long Term Effect of High Intensity Versus Low-Level Laser Therapy in Treatment of Patients With Achilles Tendinitis or Plantar Fasciitis: A Single Blinded Randomized Controlled Clinical Trial.
Brief Title: Effect of HILT vs LLLT in Treatment of Patients With Achilles Tendinitis or Plantar Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Collaborators: Research Council of Lithuania (Other)
Responsible Party: Principal Investigator, Dovile Naruseviciute, Doctor of Medicine, investigator, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-07-14 Nr.BE-2-32
Record Dates: First submitted 2019-03-03; First posted 2019-03-14 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Plantar Fascitis; Achilles Tendon Pain
Keywords: High-Intensity Laser Therapy; Low-level Laser Therapy
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants were informed that they will receive treatment with laser. Participants were not informed which laser (HILT or LLLT) was administered.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-intensity laser therapy (Experimental): The participants received stretching and exercise guidance and underwent the BTL-6000 High Intensity Laser 12 W with 10 mm pen applicator high intensity laser procedures (mode = continuous, power = 7 W, dose = 120 J/cm2, total time= 7 min. 8 sec.) 3 times per week (total of 8 procedures).
  Interventions: Device: High-intensity laser therapy
- Low-level laser therapy (Active Comparator): The participants received stretching and exercise guidance underwent the LAS-Expert with laser shower applicator Low-level Laser therapy procedures (785 nm wavelength, 4,0 J/cm2, 35cm2, 6:40 min) 3 times per week (total of 8 procedures).
  Interventions: Device: Low-level Laser therapy

INTERVENTIONS:
Device: High-intensity laser therapy — tissue photobiostimulation for pain reduction and healing enhancement.
  Other Names: BTL-6000 High Intensity Laser 12 W with 10 mm pen
  Arms: High-intensity laser therapy
Device: Low-level Laser therapy — tissue photobiostimulation for pain reduction and healing enhancement.
  Other Names: LAS-Expert with laser shower
  Arms: Low-level laser therapy

SUMMARY:
The aim of this study is to evaluate and compare the changes of heel pain, functional health and well-being after high-intensity and low-level laser therapy for plantar fasciitis or Achilles tendinopathy

DETAILED DESCRIPTION:
Plantar heel pain, also known as plantar fasciitis, causes soreness or tenderness of the sole of the foot under the heel, which sometimes extends into the medial arch. Pain associated with the condition may cause substantial disability and poor health-related quality of life. Achilles tendinitis is a common etiology of posterior heel pain that results in significant pain and loss of function. Calf exercise is initial management that may be supported by laser therapy. A treatment possibility high-intensity laser therapy is little explored. High-intensity lasers can deliver more energy deeper into tissue. The hypothesis is that both lasers are effective in treatment of plantar fasciitis or Achilles tendinopathy, but high-intensity laser therapy is more effective.

The aim of this study is to evaluate and compare the changes of heel pain, functional health and well-being after high-intensity and low-level laser therapy for plantar fasciitis or Achilles tendinopathy.

The study was approved by Committee on Biomedical Research Ethics of Kaunas Region (2016-07-14 No. BE-2-32). Patients are recruited in out patient clinic of Physical Medicine and Rehabilitation Department in The Hospital of Lithuanian University of Health Sciences (LSMU) Kauno klinikos.

ELIGIBILITY:
Inclusion Criteria:

* unilateral painful activity related symptoms from the Achilles region
* tenderness during palpation of Achilles insertion on calcaneus or couple centimeters above
* unilateral plantar heel pain, mainly during the first few steps upon rising in the morning
* tenderness at the insertion site of the plantar fascia o the calcaneus

Exclusion Criteria:

* bilateral heel pain
* other acute pathology (febrile fever, cold. etc.) that require treatment
* other painful conditions that require painkillers (tooth pain, back pain, etc)
* pregnancy
* history of recent trauma or foot surgery
* wounds, infections in treatment area
* impaired sensation in treatment area
* pigmentation changes on the skin in treatment area (tattoo, birthmarks)
* received oral or injected corticosteroids within the last 26 weeks
* diagnosis of systemic inflammatory arthritis (goat, rheumatoid arthritis, etc)
* diagnosis of neurological heel pain (radiculopathy)
* diagnosis of other heel pathology (calcaneal stress fracture, osteomyelitis, plantar fascia neoplasm, plantar fascia rupture, etc)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Pain - visual analog scale | Baseline
  Visual analog scale from 0 to 100 mm ("0" = no pain, "100" = the most intense pain). Heel pain in specific day time (at rest, first morning step, several minutes after first step, first step after prolonged sitting in the middle of the day, in the evening and at night)
Pain - visual analog scale | After 3 weeks of treatment
  Visual analog scale from 0 to 100 mm ("0" = no pain, "100" = the most intense pain). Heel pain in specific day time (at rest, first morning step, several minutes after first step, first step after prolonged sitting in the middle of the day, in the evening and at night)
Pain - visual analog scale | 4 weeks follow up
  Visual analog scale from 0 to 100 mm ("0" = no pain, "100" = the most intense pain). Heel pain in specific day time (at rest, first morning step, several minutes after first step, first step after prolonged sitting in the middle of the day, in the evening and at night)

SECONDARY OUTCOMES:
Pain - pressure algometry | Baseline to 3 weeks and 4 weeks follow up
  Pressure algometry was performed on both affected and healthy feet. It was measured with algometer (kgf)
Range of motion - goniometry | Baseline to 3 weeks and 4 weeks follow up
  Ankle and first toe dorsiflexion and plantarflexion was measured in both affected and healthy feet. It was measured in standardized position with goniometer (degrees)
Tendon thickness measurement - ultrasound | Baseline to 3 weeks and 4 weeks follow up
  Thickness of tendon was measured with ultrasound machine in longitudinal view of tendon in both affected and healthy feet (mm).
Functional health and well-being - SF-36v2® | Baseline to 3 weeks and 4 weeks follow up
  Paper questionnaire for participants to fill in. Medical Outcomes Study Short Form 36 2 version (SF-36v2) was used. Measure is divided into 8 subscales and 2 composite domains The 8 subscales are Physical Functioning, Role Limitations due to Physical Problems, General Health Perceptions, Vitality, Social Functioning, Role Limitations due to Emotional Problems, General Mental Health and Health Transition. Respondents were asked to answer items referring to the past 4 weeks Recommended scoring system for the SF-36 is a weighted Likert system for each item Items within subscales are totaled to provide a summed score for each subscale or dimension.
  Each of the 8 summed scores is linearly transformed onto a scale from 0 (negative health) to 100 (positive health) to provide a score for each subscale.
Evaluation of functional condition of patients' feet - Foot Function Index-Revised Short Form | Baseline to 3 weeks and 4 weeks follow up
  Paper questionnaire for participants to fill in. The questionnaire consists of 34 questions grouped into 5 subcategories: pain, stiffness, difficulty, activity limitation, and social issues. The answers are represented by a 4-level Likert scale. The numerical 5 is not a Likert scale; it is an option that the particular question is not applicable. A higher score represents worse condition.
Evaluation of functional condition of patients' feet - Foot and Ankle Ability Measure | Baseline to 3 weeks and 4 weeks follow up
  Paper questionnaire for participants to fill in. Foot and Ankle Ability Measure consists of the 21-item activities of daily living and 8-item Sports subscales. The response to each item is scored by Likert scale from 4 to 0, with 4 being "no difficulty" and 0 being "unable to do". A higher score represents a higher level of physical function.
Pain - numerical pain rating scale | Baseline to 3, 5, 8, 10, 12, 15 and 17 days (before every laser procedure)
  Numerical pain rating scale from 0 to 10 ("0" = no pain, "10" = the most intense pain). Heel pain in specific day time (at rest, first morning step, several minutes after first step, first step after prolonged sitting in the middle of the day, in the evening and at night)

CONTACTS AND LOCATIONS:
Overall Officials: Raimondas Kubilius, professor, Principal Investigator — Lithuanian University of Health Sciences
Locations (1):
- The Lithuanian University of Health Sciences, Department of Rehabilitation, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided